CLINICAL TRIAL: NCT05751824
Title: Evaluating the Effect of the Automatic Surveillance System on Surveillance Rate of Colorectal Postpolypectomy Patients: A Prospective, Multicenter Study
Brief Title: Evaluating the Effect of the Automatic Surveillance System on Surveillance Rate of Colorectal Postpolypectomy Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Renmin Hospital of Wuhan University (Other)
Collaborators: Jiangmen Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: EA-23-01
Record Dates: First submitted 2022-11-07; First posted 2023-03-02 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Artificial Intelligence; Surveillance
Keywords: surveillance rate; automatic surveillance
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- With automatic surveillance system (Experimental): Patients were reminded of the surveillance time by an automatic surveillance system before the surveillance time.
  Interventions: Other: AI based automatic surveillance (AS) system (ENDOANGEL-AS)
- With manual reminder (Active Comparator): Patients were reminded of the surveillance time manually before the surveillance time.
  Interventions: Other: Manually remind the patients to review.
- Normal group (No Intervention): The patients in the control group were observed in the clinical natural state of surveillance without automatic surveillance system or manual reminder.

INTERVENTIONS:
Other: AI based automatic surveillance (AS) system (ENDOANGEL-AS) — An automatic surveillance (AS) system to accurately identify post-polypectomy patients, assign surveillance intervals for different risks of patients and proactively follow up with patients at certain times.
  Arms: With automatic surveillance system
Other: Manually remind the patients to review. — Medical staff remind patients to review by telephone.
  Arms: With manual reminder

SUMMARY:
In this study, we proposed a prospective study about the effect of the automatic surveillance system on surveillance rate of colorectal postpolypectomy patients. The enrolled patients were divided into group A with intelligent surveillance system, group B with manual reminder, and group C with natural state. The surveillance among the three groups were compared.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or older who undergo colonoscopy.

Exclusion Criteria:

* 1)No pathological result.
* 2) No or invalid contact information.
* 3) The surveillance interval cannot be determined according to the surveillance guidelines, including poor bowel preparation, colorectal cancer or suspicious malignance, surgery or colorectal ESD history, those who fail to complete colonoscopy due to unbearable, pathological indications of not polyps, hamartoma or lymphoma polyps, history of ulcerative colitis, and so on.
* 4) Has participated in other clinical trials, signed the informed consent form and is in the surveillance period of other clinical trials.
* 5) Have drug or alcohol abuse or psychological disorder in the past five years.
* 6）Pregnancy.
* 7）Not suitable for recruitment after investigator evaluation because of other high-risk conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 867 (Estimated)
Dates: Start 2023-02-26 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
surveillance rate | From enrollment to study completion, assessed up to 3 years.
  The numerator is the number of patients with surveillance, and the denominator is the number of all colorectal postpolypectomy patients requiring surveillance.

SECONDARY OUTCOMES:
Advance Surveillance Rate | From enrollment to study completion, assessed up to 3 years.
  The numerator is the number of patients with surveillance in advance, and the denominator is the number of all colorectal postpolypectomy patients requiring surveillance.
On-time Surveillance Rate | From enrollment to study completion, assessed up to 3 years.
  The numerator is the number of patients with on-time surveillance, and the denominator is the number of all colorectal postpolypectomy patients requiring surveillance.
Delayed Surveillance Rate | From enrollment to study completion, assessed up to 3 years.
  The numerator is the number of patients with delayed surveillance, and the denominator is the number of all colorectal postpolypectomy patients requiring surveillance.
The accuracy of identifing post-polypectomy patients | At the time of enrollment.
  The numerator is the number of patients correctly identified into post-polypectomy patients, and the denominator is the number of patients undergoing colonoscopy.
The accuracy of classifying risk levels | At the time of enrollment.
  The numerator is the number of patients correctly classified by automated surveillance system, and the denominator is the number of all enrolled colorectal postpolypectomy patients.
The accuracy of assigning surveillance intervals | At the time of enrollment.
  The numerator is the number of patients correctly assigned by automated surveillance system, and the denominator is the number of all enrolled colorectal postpolypectomy patients.
lesion progression rate | From enrollment to study completion, assessed up to 3 years.
  The numerator is the number of patients with lesion progression, and the denominator is the number of all surveillance colorectal postpolypectomy patients.
lesion persistence rate | From enrollment to study completion, assessed up to 3 years.
  The numerator is the number of patients with lesion persistence, and the denominator is the number of all surveillance colorectal postpolypectomy patients.
lesion regression rate | From enrollment to study completion, assessed up to 3 years.
  The numerator is the number of patients with lesion regression, and the denominator is the number of all surveillance colorectal postpolypectomy patients.
The incidence rate of colorectal cancer | From enrollment to study completion, assessed up to 3 years.
  The numerator is the number of patients with colorectal cancer in surveillance colonoscopy, and the denominator is the number of all surveillance colorectal postpolypectomy patients.

CONTACTS AND LOCATIONS:
Overall Officials: Honggang Yu, phD, Principal Investigator — Renmin Hospital of Wuhan University
Locations (2):
- China (2):
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Renmin Hospital of Wuhan University, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No